CLINICAL TRIAL: NCT03317184
Title: Hand-Assisted Laparoscopic Donor Nephrectomy PERiumbilical Versus Pfannenstiel Incision and Return to Normal Physical ACTivity: A Randomized Clinical Trial: HAPERPACT Trial
Brief Title: Hand-assisted Laparoscopic Donor Nephrectomy Periumbilical Versus Pfannenstiel Incision
Acronym: HAPERPACT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Heidelberg (Other)
Responsible Party: Principal Investigator, Dr. A. Mehrabi, MD, University Hospital Heidelberg
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: S-291/2017
Record Dates: First submitted 2017-10-06; First posted 2017-10-23 (Actual); Last update posted 2018-05-14 (Actual); Status verified 2018-05

CONDITIONS: Donor Nephrectomy
Keywords: Physical Activity; Pfannenstiel incision; Periumbilical incision
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: Expertise-based, single intuition, assessor-blinded, randomized clinical trial.
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Periumbilical incisions (Experimental)
  Interventions: Procedure: Periumbilical incision
- Pfannenstiel incision (Experimental)
  Interventions: Procedure: Pfannenstiel incision

INTERVENTIONS:
Procedure: Periumbilical incision — A periumbilical incision is made at the abdominal midline for hand-assisted laparoscopic donor nephrectomy.
  Arms: Periumbilical incisions
Procedure: Pfannenstiel incision — Pfannenstiel incision is made as a slightly curved horizontal line just above the pubic symphysis for hand-assisted laparoscopic donor nephrectomy.
  Arms: Pfannenstiel incision

SUMMARY:
Despite efforts to optimize the transplantation of deceased donor kidneys, the number of available kidneys continues to fall short of the demand. Living donor kidneys have been used to overcome this shortage. Graft and patient survival is significantly higher following living donor kidney transplantation compared with deceased donor kidney transplantation. Open donor nephrectomy was the universal technique prior to the advent of laparoscopic techniques. Laparoscopic approaches have definite advantages over open surgery in terms of blood loss, postoperative pain, analgesic requirements, duration of hospital stay, and convalescence. There is some controversy regarding longer warm ischemia time, longer operative time, and increased bleeding with laparoscopic nephrectomy compared with hand-assisted laparoscopic living donor nephrectomy (HALDN). HALDN attempted to reduce warm ischemia time by using the hand port to extract the kidney instantly after dividing the blood vessels. This technique also offers tactile feedback, better manual control of bleeding, a relatively shorter learning curve, less kidney traction, faster kidney removal, and shorter warm ischemic periods. HALDN is often performed using periumbilical and Pfannenstiel incisions for hand-assisted port placement. Pfannenstiel incisions improve wound complications such as incisional hernia, cosmetic issues, and wound dehiscence. However, duration of surgery, postoperative pain score, and length of hospital stay are significantly lower in donors with periumbilical incisions.To the best of our knowledge, these two types of incision have not been compared in a randomized controlled trial in patients undergoing HALDN. Our objective is to compare the results of Pfannenstiel incision (intervention group) with periumbilical incision (control group). The return to normal physical activity will be evaluated in a clinical randomized trial using an expertise-based design.

DETAILED DESCRIPTION:
Despite all efforts to optimize the transplantation of deceased donor kidneys, the number of available kidneys continues to fall short of demand. Living donor kidneys have been used to overcome this organ shortage. Graft and patient survival is significantly higher following living donor kidney transplantation compared with deceased donor kidney Transplantation.

The major disadvantage of using living donors is that a healthy individual must undergo a major surgical procedure to provide the organ for transplantation. The donor does not medically benefit from the procedure, but there is a medical impact on both donor and recipient. Therefore, a nephrectomy technique associated with the lowest donor risk and the best organ quality should be used during Transplantation.

Open donor nephrectomy was the universal technique before the advent of laparoscopic techniques. Laparoscopic living donor nephrectomy was introduced in 1995 and commercial ports were developed shortly after. In 1998, Wolf et al. described the hand-assisted laparoscopic living donor nephrectomy (HALDN) technique and since then it has become widely adopted. Laparoscopic methods have definite advantages over open surgery in terms of blood loss, postoperative pain, analgesic requirements, duration of hospital stay, and convalescence.

There is some controversy regarding the possibility of relatively longer warm ischemia time, longer operative time, and increased bleeding with laparoscopic nephrectomy. HALDN reduces warm ischemia time by extracting the kidney using the hand port as soon as the blood vessels are divided. This technique is associated with tactile feedback, better manual control of bleeding, relatively shorter learning curve, less kidney traction, faster kidney removal, and shorter warm ischemic periods. At present, there is no strong evidence to support the use of one laparoscopic approach in preference to the other. However, evidence suggests that HALDN is the most cost-effective method of donor surgery and achieves equivalent clinical benefits of pure laparoscopic approaches with less operative time.

HALDN is usually performed using a periumbilical or Pfannenstiel incision for hand-assisted port placement and kidney extraction. A periumbilical incision is made at the midline. In contrast, a Pfannenstiel incision is made as a slightly curved horizontal line just above the pubic symphysis. Pfannenstiel incisions improve wound complications, such as incisional hernia, cosmetic results, and wound dehiscence. However, the duration of surgery, postoperative pain score, and length of hospital stay were significantly lower in donors with periumbilical incision. The inserted hand plays a vital role in the procedure, including retraction and dissection, therefore the hand port midline incision is placed close to the periumbilical area. Dissecting the upper pole of the kidney through a Pfannenstiel incision may be difficult in morbidly obese and large donors.

Patients with Pfannenstiel incisions return to normal physical activity quicker than those with periumbilical incisions. However, to the best of our knowledge, these two different incision types in patients undergoing HALDN have not been compared in a randomized controlled trial.Our objective is to compare the return of patients to physical activity following a HALDN procedure with Pfannenstiel incision (intervention group) or periumbilical incision (control group) in a clinical randomized trial using an expertise-based design.

ELIGIBILITY:
Inclusion Criteria:

* Age > 20 years
* No permanent pain therapy
* Kidneys with only a single artery and vein in the graft
* Informed consent for participation provided

Exclusion Criteria:

* Infection or scar present precluding incision placement at one of the randomization sites
* Bleeding disorders
* Chronic use of immunosuppressive agents (e.g. steroids)

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2017-11-01 (Actual); Primary Completion 2020-02-01 (Estimated); Study Completion 2020-06-01 (Estimated)

PRIMARY OUTCOMES:
Days to return to normal physical activity | Four weeks
  Patients will be asked to complete the "Katz basic activities of daily living" self-maintenance questionnaire each day for 4 weeks after the operation. This questionnaire assesses the ability to perform daily living activities (0 = no activity and 6 = normal activity). The normal physical activity is perceived as good.

SECONDARY OUTCOMES:
Warm ischemia time | One day
  From the time of clamping of the first renal artery in situ to flushing of the kidney with chilled solution on the back table
Intraoperative complications | One day
  From skin incision to skin closure
Estimated blood loss | One day
  From skin incision to skin closure
Operating time | One day
  From skin incision to skin closure
Postoperative pain | Seven days
  Severity of pain via 11-point Visual Analogue Scale (0 = no pain and 10 = unbearable distress).
Rescue analgesic | Seven days
  Total amount of analgesics required.
Peak expiratory flow rate | Seven days
  Is defined as maximum speed of expiration, as measured with a peak flow meter.
Postoperative complications | 60 days
  According to the Clavien-Dindo classification
Length of hospital stay | 60 days
  From the day of the operation until the day of discharge
Time to return to work | 60 days
  From the day of discharge and return to work
Physical activity score | 60 days
  The International Physical Activity Questionnaire, Short Form (IPAQ) will be used as an indicator of physical activity and fitness. IPAQ assesses total physical activity in the previous 7 days. Questions measure the frequency (days per week) and duration (minutes per session) of physical activity, as well as its intensity level (vigorous, moderate, walking, or sitting). Participants are categorized into one of three physical activity levels (low, moderate, high). Range is not applicable because it is a categorical variable. The high activity category is perceived as good.
Patient satisfaction | 60 days
  Patient satisfaction score via 5-point Likert scale (5 = representing strongly satisfied and 1 = representing strongly unsatisfied).
Cosmetic score | 60 days
  As defined by the Stony Brook scar scale (SBSES). The SBSES assessed five scar components: width, height, color, suture marks and overall appearance. Each component was assigned a score of 0 or 1 with a total sum range of 0 (worst) to 5 (best).
Incisional hernia | 60 days
  Defined as a fascia or muscle defect (bulging hernial sac and palpable fascia gap) at the site of the surgical incision examined by palpation and ultrasonography.
Mortality | 60 days
  Death due to any cause.
Recipient serum creatinine level | 30 days
  Serum creatinine level (mg/dL)
Glomerular filtration rate | 30 days
  GFR (mL/min/1.73 m2) calculated with "175 × (Scr)-1.154 × (Age)-0.203 × (0.742 if female)" Formula
Delayed graft function | 30 days
  Is defined as the need for one or more hemodialysis treatments following transplantation prior to the onset of graft function.
Primary non-function | 30 days
  A recipient whose graft never functions.

CONTACTS AND LOCATIONS:
Overall Officials: Yakup Kulu, MD, Principal Investigator — Department of General, Visceral and Transplant Surgery, University Hospital Heidelberg, Germany; Arianeb Mehrabi, MD, Study Director — Department of General, Visceral and Transplant Surgery, University Hospital Heidelberg, Germany
Locations (1):
- Division of Visceral Transplantation, Department of General, Visceral and Transplantation Surgery, University of Heidelberg, Heidelberg, Baden-Wurttemberg, Germany

REFERENCES:
- [Derived] Kulu Y, Muller-Stich BP, Ghamarnejad O, Khajeh E, Polychronidis G, Golriz M, Nickel F, Benner L, Knebel P, Diener M, Morath C, Zeier M, Buchler MW, Mehrabi A. Hand-Assisted laparoscopic donor nephrectomy PERiumbilical versus Pfannenstiel incision and return to normal physical ACTivity (HAPERPACT): study protocol for a randomized controlled trial. Trials. 2018 Jul 13;19(1):377. doi: 10.1186/s13063-018-2775-4. PMID 30005640